CLINICAL TRIAL: NCT06771635
Title: Effects of a Targeted Concurrent Training Program on the Exercise Adherence in Female Breast Cancer Survivors: a Randomized Controlled Trial
Brief Title: Effect of Physical Training Program on the Exercise Adherence for Breast Cancer Survivor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Burgos (Other)
Collaborators: Fundación Instituto Valenciano de Oncología (Other); Fundación Trinidad Alfonso (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2018/0009
Record Dates: First submitted 2025-01-07; First posted 2025-01-13 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer Stage I; Breast Cancer Stage II; Breast Cancer Stage III; Breast Cancer Stage IIIA
Keywords: Breast Cancer; Physical activity; Adherence; Concurrent training
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: Is a prospective, multicenter, randomized, parallel-controlled, prospective pilot study
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Concurrent Training Program (Experimental): This group will participate in a 6-week concurrent training program.
  Interventions: Other: concurrent
- Health Education Only (Control) (Active Comparator): This group will no participate in the concurrent training intervention program.
  Interventions: Behavioral: Health Education Session

INTERVENTIONS:
Other: concurrent — The concurrent training program is divided into three types of training: endurance, cardiovascular and neuromotor.
  Resistance training sessions were performed in a circuit format with >30" rest periods between exercises. The volume of work ranged from 8 to 12 repetitions at 60% of the estimated 1 maximum repetition (RM).
  The cardiovascular work time per session ranged from 25-50 min depending on the intensity of the exercise and the intensity was regulated according to the maximum heart rate (FHR) estimated for each subject between 60-75%
  The neuromotor training intensity of the sessions was low. The participants wore a heart rate monitor and were instructed not to exceed 60% of their HRF
  Arms: Concurrent Training Program
Behavioral: Health Education Session — Single formative session on healthy lifestyle and nutrition provided to both groups. Control group received only this session without concurrent training.
  Arms: Health Education Only (Control)

SUMMARY:
Breast cancer (BC) is one of the most common cancers among women worldwide, with survival rates steadily improving due to advances in early detection and treatment. Despite these improvements, survivors frequently experience long-term side effects such as fatigue, reduced physical function, osteosarcopenia (loss of muscle mass and bone density), and diminished quality of life (QOL). These sequelae often lead to loss of independence, increased frailty, and reduced participation in daily activities. Physical activity, particularly structured and supervised programs, has been shown to mitigate many of these effects. Concurrent training, which combines strength, cardiovascular, and neuromotor exercise, provides a comprehensive approach that targets muscle mass, bone health, and functional mobility. However, adherence to regular physical activity in this population remains low, with most survivors not achieving recommended levels of at least 150 minutes per week of moderate-to-vigorous exercise. This pilot randomized controlled trial aims to evaluate the effects of a 6-week supervised concurrent training program in breast cancer survivors. The program includes 12 supervised sessions designed to improve exercise adherence, physical activity levels, and QOL. The intervention is compared with a control group that receives only a health education session. Outcomes include QOL assessed by the FACT-B questionnaire, physical activity levels measured by the GPAQ, sedentary time, functional fitness, anthropometry, and patient satisfaction. The study is expected to provide evidence that a short-term supervised concurrent training program can improve emotional well-being, preserve QOL, and increase adherence to physical activity in breast cancer survivors.

DETAILED DESCRIPTION:
This randomized, multicenter, parallel-controlled pilot trial was conducted in two tertiary hospitals in Spain to evaluate the effects of a short-term supervised concurrent training program on physical activity adherence and quality of life in breast cancer survivors.

Participants allocated to the intervention group completed a 6-week supervised concurrent training program consisting of 12 sessions (two sessions per week, approximately 60 minutes per session). The training program combined resistance, cardiovascular, and neuromotor exercises and was designed to address muscle strength, cardiorespiratory fitness, coordination, and functional mobility. Exercise sessions were supervised by qualified exercise professionals trained in oncology rehabilitation. Exercise intensity was individually adjusted and monitored to ensure participant safety and adherence to the prescribed training load.

The control group attended a single educational session focused on healthy lifestyle and nutrition and did not participate in the exercise program. Both groups continued to receive usual oncological follow-up throughout the study period.

Assessments were conducted at baseline, immediately after the intervention (6 weeks), and during follow-up at 3 and 6 months to evaluate changes over time. Ethical approval was obtained from the institutional ethics committees of the participating centers (protocol code 2018/0009), and written informed consent was obtained from all participants prior to study participation.

ELIGIBILITY:
Inclusion Criteria:

* Stage I-IIIA
* Free of disease
* Without active chemotherapeutic treatment

Exclusion Criteria:

* Patients suffered from a chronic disease that prevented them from physical activity program
* Patients with sequelae of surgery, edema of >2 degrees in extremities with lymphadenectomy
* Those women who performed PA according to the recommendations established by the WHO.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2019-04-08 (Actual); Study Completion 2019-07-19 (Actual)

PRIMARY OUTCOMES:
Change in Quality of Life (Functional Assessment of Cancer Therapy-Breast [FACT-B] Total Score) | Baseline, post-intervention (6 weeks), 3 months, and 6 months.
  Quality of life assessed using the Functional Assessment of Cancer Therapy-Breast (FACT-B) questionnaire. The FACT-B total score ranges from 0 to 148 points, with higher scores indicating better quality of life.

SECONDARY OUTCOMES:
Change in Emotional Well-Being (Functional Assessment of Cancer Therapy-Breast Emotional Well-Being Subscale) | Baseline, post-intervention (6 weeks), 3 months, and 6 months.
  Emotional well-being assessed using the Emotional Well-Being subscale of the Functional Assessment of Cancer Therapy-Breast (FACT-B) questionnaire. The subscale score ranges from 0 to 24 points, with higher scores indicating better emotional well-being.
Change in Physical Activity Level (MET-min/week, GPAQ) | Baseline, post-intervention (6 weeks), 3 months, and 6 months.
  Physical activity levels assessed using the Global Physical Activity Questionnaire (GPAQ). Data expressed in MET-minutes per week across work, transport, and leisure domains.
Mean Sedentary Time (minutes/day, GPAQ) | Baseline, post-intervention (6 weeks), 3 months, and 6 months.
  Sedentary behavior measured using the GPAQ. Time spent sitting or reclining per day is recorded in minutes.
Adherence to Exercise Program (percent of sessions attended) | During the 6-week intervention period.
  Exercise adherence calculated as the percent of supervised exercise sessions attended out of the 12 prescribed sessions during the intervention period
Change in Weight (kg) | Baseline, post-intervention (6 weeks), 3 months, and 6 months
  Body weight measured with a calibrated SECA® scale.
Change in Height (cm) | Baseline, post-intervention (6 weeks), 3 months, and 6 months.
  Height measured with a stadiometer.
Change in Body Mass Index (kg/m²) | Baseline, post-intervention (6 weeks), 3 months, and 6 months.
  Body mass index calculated as weight (kg)/height (m²).
Change in Handgrip Strength (kg, dynamometer) | Baseline, post-intervention (6 weeks), 3 months, and 6 months.
  Handgrip strength measured using a handheld dynamometer, following standardized ACSM protocols.
Change in Cardiorespiratory Fitness (Harvard Step Test Fitness Index) | Baseline, post-intervention (6 weeks), 3 months, and 6 months.
  Cardiorespiratory fitness assessed using the Harvard Step Test Fitness Index, which typically ranges from 0 to 150 units, with higher scores indicating better cardiorespiratory fitness.
Patient Satisfaction with the Intervention (Study-Specific Satisfaction Questionnaire) | Immediately post-intervention (6 weeks).
  Patient satisfaction assessed using a study-specific satisfaction questionnaire scored on a 0 to 5 Likert scale, where 0 indicates very dissatisfied and 5 indicates very satisfied. Higher scores indicate greater satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Mielgo-Ayuso, PhD, Study Director — Universidad de Burgos
Locations (1):
- Universidad de Burgos, Burgos, Burgos, Spain

IPD SHARING:
Plan to Share IPD: No
Only IPD used in the results publication

REFERENCES:
- [Result] Cao C, Friedenreich CM, Yang L. Association of Daily Sitting Time and Leisure-Time Physical Activity With Survival Among US Cancer Survivors. JAMA Oncol. 2022 Mar 1;8(3):395-403. doi: 10.1001/jamaoncol.2021.6590. PMID 34989765
- [Result] Weiner LS, Takemoto M, Godbole S, Nelson SH, Natarajan L, Sears DD, Hartman SJ. Breast cancer survivors reduce accelerometer-measured sedentary time in an exercise intervention. J Cancer Surviv. 2019 Jun;13(3):468-476. doi: 10.1007/s11764-019-00768-8. Epub 2019 May 29. PMID 31144265
- [Result] Friedenreich CM, Cust AE. Physical activity and breast cancer risk: impact of timing, type and dose of activity and population subgroup effects. Br J Sports Med. 2008 Aug;42(8):636-47. doi: 10.1136/bjsm.2006.029132. Epub 2008 May 16. PMID 18487249